CLINICAL TRIAL: NCT02803372
Title: Impact of Circulatory Management Based on LiDCOrapid Hemodynamic Monitoring on the Incidence of Acute Kidney Injury in Patients Undergoing Partial Nephrectomy: A Randomized Controlled Trial
Brief Title: Circulatory Management and Acute Kidney Injury in Patients Undergoing Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016[1118]
Record Dates: First submitted 2016-06-06; First posted 2016-06-17 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Acute Kidney Injury
Keywords: partial nephrectomy; acute kidney injury; LiDCOrapid; circulatory management
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): In addition to routine monitoring, invasive LiDCOrapid is used to monitor mean arterial pressure (MAP), stroke volume variation (SVV) and cardiac index (CI). Intraoperative goal-directed circulatory management is performed, i.e., to maintain MAP > 95 mmHg, SVV < 6%, and CI 3.0-4.0 L/min/m2, started from renal artery clamping and maintained until the end of surgery.
  Interventions: Other: Goal-directed circulatory management
- Control group (Active Comparator): Routine monitoring is performed, which includes invasive blood pressure and urine output. Intraoperative routine circulatory management is performed, i.e., to maintain blood pressure within 20% from baseline level and urine output > 0.5 ml/kg/h.
  Interventions: Other: Routine circulatory management

INTERVENTIONS:
Other: Goal-directed circulatory management — In addition to routine monitoring, invasive LiDCOrapid is used to monitor MAP, SVV and CI. Intraoperative circulatory management is performed according to the goal-directed principal, i.e., to maintain MAP > 95 mmHg, SVV < 6%, and CI 3.0-4.0 L/min/m2, started from renal artery clamping and maintained until the end of surgery. Crystalloid solution is firstly infused to maintain SVV at the target level, dobutamine and/or noradrenaline are then infused to maintain MAP and CI at the target levels.
  Arms: Intervention group
Other: Routine circulatory management — Routine monitoring is performed, which include invasive blood pressure and urine output. Intraoperative circulatory management is performed according to routine practice, i.e., to maintain blood pressure within 20% from baseline level and urine output > 0.5 ml/kg/h by infusing crystalloid solution and administering vasoactive drugs when considered necessary.
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate whether circulatory management based on LiDCOrapid hemodynamic monitoring can reduce the incidence of acute kidney injury in patients undergoing partial nephrectomy when compared with routine circulatory management based on blood pressure and urine output monitoring

DETAILED DESCRIPTION:
Previous studies found that the incidence of acute kidney injury afer partial nephrectomy is higher than 30%. In addition to nephron loss induced by renal parenchyma resection, ischemia/reperfusion injury produced by clamping/unclamping of renal arteries is also an important reason. However, studies investigating the effect of circulatory management on the incidence of acute kidney injury after partial nephrectomy are limited.

It has been shown that perioperative hemodynamic optimization protected renal function in surgical patients. And in patients undergoing renal transplantation, adequate hydration and optimal perfusion enhances early graft function. The investigators hypothesize that hydration and circulatory management to guarantee optimal renal perfusion may decrease the occurrence of acute kidney injury after partial nephrectomy. The purpose of this study is to investigate whether circulatory management based on LiDCOrapid hemodynamic monitoring can reduce the incidence of acute kidney injury in patients undergoing partial nephrectomy when compared with routine circulatory management based on blood pressure and urine output monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Planning to undergo partial nephrectomy;

Exclusion Criteria:

1. Patients with renal function damage (chronic kidney disease stage 3-5) before surgery;
2. Patients with arrhythmia or aortic valve diseases (moderate or higher degree stenosis/regurgitation);
3. Patients who has participated in other trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury after surgery | During the first 3 days after surgery
  Acute kidney injury is diagnosed according to KDIGO (Kidney Disease: Improving Global Outcomes) criteria

SECONDARY OUTCOMES:
Serum creatinine concentration | At 3 and 6 months after surgery
  Serum creatinine concentration
Length of stay in hospital after surgery | From end of surgery to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of postoperative complications | From end of surgery to 30 days after surgery
  Incidence of complications within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data of individual participants for all primary and secondary outcome measures will be made available on request after study completion and paper publication.

REFERENCES:
- [Background] Rajan S, Babazade R, Govindarajan SR, Pal R, You J, Mascha EJ, Khanna A, Yang M, Marcano FD, Singh AK, Kaouk J, Turan A. Perioperative factors associated with acute kidney injury after partial nephrectomy. Br J Anaesth. 2016 Jan;116(1):70-6. doi: 10.1093/bja/aev416. PMID 26675951
- [Background] De Gasperi A, Narcisi S, Mazza E, Bettinelli L, Pavani M, Perrone L, Grugni C, Corti A. Perioperative fluid management in kidney transplantation: is volume overload still mandatory for graft function? Transplant Proc. 2006 Apr;38(3):807-9. doi: 10.1016/j.transproceed.2006.01.072. PMID 16647477
- [Background] Aulakh NK, Garg K, Bose A, Aulakh BS, Chahal HS, Aulakh GS. Influence of hemodynamics and intra-operative hydration on biochemical outcome of renal transplant recipients. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):174-9. doi: 10.4103/0970-9185.155144. PMID 25948896
- [Background] O'Loughlin E, Ward M, Crossley A, Hughes R, Bremner AP, Corcoran T. Evaluation of the utility of the Vigileo FloTrac() , LiDCO() , USCOM and CardioQ() to detect hypovolaemia in conscious volunteers: a proof of concept study. Anaesthesia. 2015 Feb;70(2):142-9. doi: 10.1111/anae.12949. PMID 25583188
- [Background] Chin JH, Jun IG, Lee J, Seo H, Hwang GS, Kim YK. Can stroke volume variation be an alternative to central venous pressure in patients undergoing kidney transplantation? Transplant Proc. 2014 Dec;46(10):3363-6. doi: 10.1016/j.transproceed.2014.09.097. PMID 25498052
- [Derived] Wu QF, Kong H, Xu ZZ, Li HJ, Mu DL, Wang DX. Impact of goal-directed hemodynamic management on the incidence of acute kidney injury in patients undergoing partial nephrectomy: a pilot randomized controlled trial. BMC Anesthesiol. 2021 Mar 3;21(1):67. doi: 10.1186/s12871-021-01288-8. PMID 33658007